CLINICAL TRIAL: NCT07371572
Title: The Efficacy and Safety of Intramuscular Methylprednisolone in Patients With Hand OsteoArthritis - the IMHOA Trial
Brief Title: The Efficacy and Safety of Intramuscular Methylprednisolone in Patients With Hand OsteoArthritis
Acronym: IMHOA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sint Maartenskliniek (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025.03; 2024-518344-20-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-22; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-09

CONDITIONS: Hand Osteoarthritis
MeSH Terms: interventions — Methylprednisolone Acetate; Methylprednisolone; Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: The first phase of the trial will include a parallel interventional study model. In the second phase, all participants will receive the same intervention (120mg methylprednisolone) on demand, which will explain as the single group model.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 120mg (Experimental): 120mg methylprednisolone acetate (3ml)
  Interventions: Drug: 120mg methylprednisolone acetate
- 40mg (Experimental): 40mg methylprednisolone acetate (1ml + 2 ml NaCl 0.9%)
  Interventions: Drug: 40mg methylprednisolone acetate
- Placebo (Placebo Comparator): Placebo (3ml NaCl 0.9%)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 120mg methylprednisolone acetate — One single intramuscular injection with 120mg methylprednisolone will be administered at baseline to each participant in the first phase.
  During the second phase, participants may receive intramuscular methylprednisolone on demand at the dosage of 120mg only if they fulfil the following conditions: hand pain >30mm on a VAS (0-100mm) and a minimum of 16 weeks interval between two consecutive injections.
  Other Names: Depo-medrol; Medrol Acetate; Depo-Medrone
  Arms: 120mg
Drug: 40mg methylprednisolone acetate — One single intramuscular injection with 40mg methylprednisolone will be administered at baseline to each participant in the first phase.
  Other Names: Medrol Acetate; Depo-Medron; Depo-Medrol
  Arms: 40mg
Drug: Placebo — One single intramuscular injection of placebo (NaCl 0.9%) will be administered at baseline to each participant in this phase.
  Other Names: 0.9% NaCl; sodium chloride 0.9%
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to determine the efficacy and safety of intramuscular methylprednisolone in patients with hand osteoarthritis. The main question it aims to answer is what the difference is in hand pain 4 weeks after the first injection with methylplrednisolone. This main goal will be assessed in the first 16 weeks, the RCT phase. Researchers will compare 120mg methylprednisolone with 40mg methylprednisolone and placebo to see if there is a difference in hand pain after 4 weeks.

Participants will be asked to visit the hospital for:

* injection of the study material
* ultrasound assessment
* physical examination like joint assessments and grip strenght
* examination of blood
* x-ray of the hand

In phase 2, from week 16 to 48, an open label phase focusing on treatment strategy and safety. In this phase all participants may receive intramuscular methylprednisolone on demand at the dosage of 120mg only if they fulfil the following conditions: hand pain > 30mm on a VAS (0-100mm) and a minimum of 16 weeks interval between two consecutive injections. Therefore, a maximum of two injections could be received during this period. Irrespective of that, all participants will be followed-up until week 48 when the end-of-study visit will take place.

ELIGIBILITY:
Inclusion Criteria:

* Patients with interphalangeal hand OA (according to the EULAR classification criteria 2023) based on patient report (age, morning stiffness) and radiographs of ≤6 months old (osteophytes, JSN (joint space narrowing) and symptom-structure concordance (present if majority (≥50%) of the symptomatic joints demonstrate radiographic findings)).
* Age ≥ 16 years
* Have hand pain >40mm on a 100mm visual analogue scale (VAS)
* Have previously experienced failure of at least one conventional type of pain medication, (self-reported of insufficient effect from topical or oral NSAID, etc. with exclusion of paracetamol)

Exclusion Criteria:

* Comorbidity

  * Chronic inflammatory (rheumatic) diseases
  * Infectious diseases
  * Known Osteoporosis
  * Known Diabetes
  * Previous diagnosis of fibromyalgia
  * Known myasthenia gravis
* Previous surgical interventions on the hand (e.g. carpal tunnel syndrome, etc.)
* Use of other Medication: In order to maximize the generalizability of the study interactions between methylprednisolone and co-medication is only prohibited when the Dutch Medication Surveillance System (Z-index) gives a signal for this interaction.
* Patients with a contraindication for MP

  * Current Gastric and duodenal ulcers
  * Current infections
  * Liver cirrhosis
  * Pregnant or breastfeeding
  * Known non-response or intolerance for MP
* Not able to read or write the Dutch language
* Neurological diagnosis

  * Epilepsy
  * Risk of psychiatric disorder

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2025-10-28 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Efficacy of intramuscular methylprednisolone acetate in reducing hand pain between baseline and week 4, compared to placebo measured on a 0-100 mm Visual Analogue Scale | From baseline to week 4
  The primary objective of this study is to assess the efficacy of intramuscular methylprednisolone acetate (120mg or 40mg) in reducing hand pain between baseline and week 4, compared to placebo measured on a digital Visual Analogue Scale ranging from 1-100 mm. The higher the score, the worse the outcome.

SECONDARY OUTCOMES:
Non-inferiority of 40mg compared to 120mg MP of the efficacy of intramuscular methylprednisolone acetate in reducing hand pain assessed by the digital 0-100 mm Visual Analogue Scale | From baseline to week 4
  Investigate non-inferiority of 40mg MP compared to 120mg MP (in case superiority to placebo of both interventions is proven in the primary analysis) of the efficacy of intramuscular methylprednisolone acetate in reducing hand pain measured on a digital Visual Analogue Scale ranging from 1-100 mm. The higher the score, the worse the outcome.
Change in hand pain at week 4, and thereafter every 4 weeks | From week 8 to week 48
  Compare the three treatment arms based on change in hand pain at week 8, and therafter every 4 weeks until week 48 measured on a digital Visual Analogue Scale ranging from 1-100 mm. The higher the score, the worse the outcome.
Percentage of participants with a reduction in hand pain larger than the MCID | From baseline to week 4
  Compare the three treatment arms based on percentage of participants with a reduction in hand pain larger than the minimal clinically important difference in pain (MCID) = 10 mm
Hand function, change in functional index | From baseline to week 48
  Compare the three treatment arms based on hand function. Change in functional index for hand OA at week 4, 16, 32 and 48, compared to baseline measured with Michigan Hand outcomes Questionnaire ranging from 0-100. The higher the score, the better the hand function.
OMERACT-OARSI responder criteria based on pain measured with Visual Analogue Scale | From baseline to week 48
  Compare the three treatment arms based on OMERACT-OARSI responder criteria based on pain measured on a digital Visual Analogue Scale ranging from 1-100 mm. The higher the score, the worse the outcome. Proportion participants fulfilling responder criteria every 4 weeks compared to baseline.
OMERACT-OARSI responder criteria based on Visual Analogue Scale hand function | From baseline to week 48
  Compare the three treatment arms based on OMERACT-OARSI responder criteria based on hand function measured on a digital Visual Analogue Scale ranging from 1-100 mm. The higher the score, the worse the outcome. Proportion participants fulfilling responder criteria every 4 weeks compared to baseline.
OMERACT-OARSI responder criteria based on patient global assessment measured with Visual Analogue Scale | From baseline to week 48
  Compare the three treatment arms based on OMERACT-OARSI responder criteria based on patient global assessment measured on a digital Visual Analogue Scale ranging from 1-100 mm. The higher the score, the worse the outcome. Proportion participants fulfilling responder criteria every 4 weeks compared to baseline.
Quality of life, measured with EuroQuol-5D-5L | From baseline to week 48
  Compare the three treatment arms based on Quality of Life, measured with EuroQuol-5D-5L questionnaire at week 16, 32 and 48.
  The EuroQol EQ-5D-5L has two measurement systems: the health state index score and the EQ Visual Analogue Scale (EQ VAS). The health state index score ranges from below zero to 1, with 1 being full health and values below zero indicating a state worse than death, depending on the specific country's value set. The EQ VAS, which measures current overall health, ranges from 0 to 100, where 100 is the best imaginable health
Patient experience of steroid use with the Steroid PRO | From baseline to week 48
  Compare the three treatment arms based on patient experience of steroid use with the Steroid PRO questionnaire every 4 weeks. Answers can be ranged from 1 to 5. Where the higher the score, the worse the outcome.
Changes in local inflammation of hand joints, determined with ultrasound | From baseline to week 4
  Compare the three treatment arms based on changes in local inflammation of the hand joints, determined with Ultrasound (US). US of hands to assess change in DIP/PIP joints at week 4 compared to baseline with change in power doppler and Greyscale score. Scores of effusion, proliferation, osteophytes and power doppler are scored between 0 to 3, where the higher the score, the worse the outcome.
Structural changes based on X-ray of the hands | From baseline to week 48
  Compare the three treatment arms based on structural changes based on X-ray of the hands to determine joint space narrowing, erosive or non-erosive, DIP/PIP joints and osteophytes between baseline and 48 weeks follow-up.
Effect on joints based on swollen joint count and tender joint count | From baseline to week 48
  Compare the three treatment arms based on effect on affected joints based on swollen joint count (SJC) and tender joint count (TJC) at baseline, week 4 and week 48.
Changes of systemic inflammation | From baseline to week 48
  Compare the three treatment arms based on changes of systemic inflammation assessed by C-reactive protein (CRP) at week 4, 16, and 48 compared to baseline. This is scored as: normal levels being less than 10 mg/L or less than 1 mg/dL. Mild elevations (10-40 mg/L) often indicate mild infection or chronic conditions, while high levels (>40 mg/L) suggest more significant inflammation, acute bacterial infection, or autoimmune disease.
Changes of systemic inflammation | From baseline to week 48
  Compare the three treatment arms based on changes of systemic inflammation assessed by Erythrocyte Sedimentation Rate (ESR) at week 4, 16, and 48 compared to baseline. ESR can be measured in range from 0 to high levels (above 100) mm/hour. The higher the value, the worse the outcome.
Medication use, health care costs by using the iMTA Productivity Cost Questionnaire | From baseline to week 48
  Compare the three treatment arms based on medication use, health care use and costs by using the iMTA Productivity Cost Questionnaire (iPCQ). It measures health-related productivity losses in the form of monetary values rather than standard units of measurement. It collects data on absenteeism and presenteeism in paid work and productivity loss in unpaid work, which is then used to calculate productivity costs in a currency.
Medication use, health care costs by using the iMTA Medical Consumption Questionnaire | From baseline to week 48
  Compare the three treatment arms based on medication use, health care use and costs by using the iMTA Medical Consumption Questionnaire (iMCQ). The iMCQ is an instrument for measuring medical consumption. The iMCQ includes questions related to frequently occurring contacts with health care providers.
Explore correlation of baseline values within treatment reponse and develop prediction model | From baseline to week 48
  Correlation between baseline clinical and imaging measures - pain severity (VAS, 0-100 mm), hand function (VAS score, 0-100 mm), grip strength (kg, dynamometer), and synovitis (ultrasound, 0-3 scale) - and treatment response, defined by the OMERACT-OARSI responder criteria (% of patients classified as responders). Statistical analysis: correlation/regression and development of a multivariable prediction model.
Explore subgroups according to structural changes on X-ray of the hand based on erosive or non-erosive, DIP osteophytes or PIP osteophytes, DIP joint space narrowing or PIP joint space narrowing at baseline. | From baseline to week 48
  Explore subgroups according to structural changes on X-ray of the hand based on erosive or non-erosive, DIP osteophytes or PIP osteophytes, DIP joint space narrowing or PIP joint space narrowing at baseline.
Assess safety of methylprednisolone 120mg or 40mg compared to placebo by assessing incidence density and cumulative incidence of AEs and SAEs | From baseline to week 48
  Assess the safety of methylprednisolone 120mg or 40mg compared to placebo by assessing incidence density and cumulative incidence of all AEs and SAEs and (S)AEs related to glucocorticoid use for each phase, using the Common Terminology Criteria for Adverse Events version 5 (CTCAEv5) and using the Glucocorticoid Toxicity Index (GTI) light.
Evaluate efficacy and safety of methylprednisolone on endpoints mentioned under 2 and 3, comparing participants based on the cumlative dose of MP | From baseline to week 48
  Evaluate efficacy and safety of methylprednisolone on endpoints mentioned under 2 and 3, comparing participants based on the cumulative dose of MP received during the study period.
Explore subgroup differences categorized by demographic factors | From baseline to week 48
  Explore subgroup differences categorized by demographic factors
Explore subgroup differences categorized by X-ray | From baseline to week 48
  Explore subgroup differences categorized by X-ray measured by joint space narrowing, osteophytes and symptom structure concordance
Explore subgroup differences categorized by ultrasound | From baseline to week 4
  Explore subgroup differences categorized by ultrasound measured by osteophytes, effusion and proliferation in DIP and PIP joints
Explore subgroup differences categorized by biomarkers in blood | From baseline to week 48
  Explore subgroup differences categorized by biomarkers in blood. Biomarkers are still unknown, and will be established during experiments.
Identification of circulating biomarkers associated with response to MP | From baseline to week 48
  Identification of circulating biomarkers associated with response to MP. Circulating biomarkers are still unknown and will be evaluated during experiments.

CONTACTS AND LOCATIONS:
Locations (1):
- Sint Maartenskliniek, Ubbergen, Gelderland, Netherlands